CLINICAL TRIAL: NCT00493584
Title: Acute Angioplasty (Primary PCI) Versus Traditional Early Invasive Treatment of Patients Presenting With NSTEMI (The Second Danish Non-ST-Elevation MI Trial - DaNSTEMI-2)
Brief Title: Acute Balloon Angioplasty vs. Traditional Early Invasive Treatment of Non-ST-Elevation Myocardial Infarction
Acronym: DaNSTEMI2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to insufficient patient inclusion the study has been stopped prematurely.
Sponsor: University of Aarhus (Other)
Collaborators: Falck Danmark (Unknown)
Responsible Party: Aarhus University Hospital, Skejby, Department of Cardiovascular research
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Thorsted 1
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Last update posted 2009-05-20 (Estimated); Status verified 2009-05

CONDITIONS: Myocardial Infarction
Keywords: Myocardial Infarction; Myocardial Ischemia; Myocardial Revascularization; Telemedicine; Percutaneous Transluminal Coronary Angioplasty
MeSH Terms: conditions — Myocardial Infarction; Myocardial Ischemia | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Primary PCI in patients with acute Non-STEMI
  Interventions: Procedure: Primary Percutaneous Coronary Intervention
- 2 (Active Comparator): Standard medical treatment and coronary angiography after 3 days in patients with Non-STEMI.
  Interventions: Procedure: Coronary angiography / Percutaneous coronary intervention

INTERVENTIONS:
Procedure: Primary Percutaneous Coronary Intervention — Coronary Angiography and PCI using standard protocols and guidelines. Contrast either Iomeron or Visipaque at the operators discretion. Equipment used for the PCI is determined at the operators discretion. All patients undergoing primary PCI receive 10.000 units of Heparin, 600 mg of Clopidogrel and a Glycoprotein IIb/IIIa inhibitor. Patients randomized to standard treatment receive 300 mg of Clopidogrel and 120IU/kg of Dalteparin b.i.d until revascularization. Glycoprotein IIb/IIIa inhibitors or thrombin inhibitors can be given as a supplement at the local hospital at the physicians discretion. All patients receive 300 mg of aspirin upon admission or diagnosis in the ambulance.
  Arms: 1
Procedure: Coronary angiography / Percutaneous coronary intervention — Coronary Angiography and PCI using standard protocols and guidelines. Contrast either Iomeron or Visipaque at the operators discretion. Equipment used for the PCI is determined at the operators discretion. All patients undergoing primary PCI receive 10.000 units of Heparin, 600 mg of Clopidogrel and a Glycoprotein IIb/IIIa inhibitor. Patients randomized to standard treatment receive 300 mg of Clopidogrel and 120IU/kg of Dalteparin b.i.d until revascularization. Glycoprotein IIb/IIIa inhibitors or thrombin inhibitors can be given as a supplement at the local hospital at the physicians discretion. All patients receive 300 mg of aspirin upon admission or diagnosis in the ambulance.
  Arms: 2

SUMMARY:
The purpose of this study is:

A) To determine whether patients with a certain type of heart attack (NSTEMI) can be reliably diagnosed in an ambulance using telemedicine. This is mandatory if NSTEMI patients in the future are to be treated with acute balloon angioplasty (primary PCI).

B) To evaluate whether primary PCI compared with the current regimen of initial medical stabilization and sub-acute PCI results in reduction of infarct-size in NSTEMI-patients.

DETAILED DESCRIPTION:
Primary PCI versus Traditional Early Invasive Treatment of Patients presenting with NSTEMI

Patients with NSTEMI are currently admitted for initial evaluation and stabilization at local hospitals. An intensive antithrombotic treatment is initiated and after 3 - 7 days of "cooling-off" the patients are referred to an invasive centre for coronary angiography and possibly PCI or CABG - this is known as the early invasive approach. Some of these patients represent a high-risk sub-group with occluded or sub-occluded coronary arteries who might benefit from very early revascularization.

Study Aims

1. To investigate if it is technically feasible to diagnose patients with NSTEMI in the pre-hospital setting and reroute them to an invasive heart centre for primary PCI in a timely manner.
2. To estimate area at risk (AAR = the part of cardiac muscle tissue at risk of infarction) and final infarct size (FIS) in patients referred for primary PCI and patients undergoing the traditional "early invasive" treatment, respectively.
3. To investigate whether Primary PCI in patients with NSTEMI results in a shorter duration of the primary admission, fewer rehospitalizations with reinfarction and acute heart failure and a briefer overall "sick leave" within a year from the index admission.

Methods

In this study 300 consecutive patients with symptoms, clinical signs and ECG changes (≥4mm cumulated or ≥ 2mm ST-segment depression (horizontal or descending) in two associated leads) suggesting significant NSTEMI are randomized for one of two strategies, either (A) usual early invasive treatment (coronary angiography and possibly PCI after 3 days) or (B) direct referral (rerouting) to primary PCI at an invasive heart centre (Skejby).

All patients undergo myocardial perfusion imaging at admission for PCI and again after 30 days to estimate AAR, FIS and possible myocardial salvage.

All patients undergo cardiac MRI on the 7th day after admission for determination of AAR and FIS.

The study is a randomized controlled study; it has been approved by the local ethics committee.

Primary outcome measures are specified above

If the study confirms that it is possible to diagnose and re-route NSTEMI patients for primary PCI with an acceptable diagnostic accuracy, then a larger scale mortality study will be planned. Furthermore, the present study will provide valuable information regarding AAR and FIS in NSTEMI-patients which may be of value for planning larger-scale, scintigraphic studies and for the possible future use of a single MRI scan to determine AAR and FIS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptoms and signs of NSTEMI and significant ECG changes (Either ≥4mm cumulated ST-segment depression (horizontal or descending), or ≥2mm ST-segment depression (horizontal or descending) in two associated leads)and/or patients with positive biomarkers for myocardial infarction (troponin T) measured in the ambulance (prehospital measurement of biomarkers).
2. Age above 18 years.
3. Tentative diagnosis made pre-hospitally.

Exclusion Criteria:

1. Severe mental or psychiatric disease (eg. psychosis, dementia, bipolar disorder or depression) as well as other conditions making it impossible to obtain informed consent.
2. Prior CABG (Coronary artery bypass graft) operation.
3. Patients with ST-depression presumed to be caused by tachycardia or cardiac hypertrophy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-03; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Final infarct size in the two study groups determined by MR | On the 7th day after admission

SECONDARY OUTCOMES:
Scintigraphic Area-At-Risk and Final-Infarct-Size in patients in group A(immediate angioplasty) and group B(early invasive strategy) respectively. | At the time of coronary angiography and after 30 days
Proportion of rerouted patients who are treated with primary PCI. | At index admission
Proportion of patients randomized to immediate angioplasty actually undergoing primary PCI within 120 minutes from first contact to health services. | At index admission
Number of readmissions in the two groups due to acute heart failure or reinfarction | 30 days and one year
Total number of days admitted at hospital in relation to the index infarction in the two groups | At index admission
Total number of days on "sick-leave" in the two groups | In relation to the index admission
Evaluation of AAR/FIS obtained by MRI on the 7th day after admission compared to AAR and FIS obtained by myocardial perfusion imaging (scintigraphy). | At the time of coronary angiography, on the 7th day after admission and after 30 days respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob T Sorensen, MD, Principal Investigator — Department of Cardiovascular research, Aarhus University Hospital, Skejby; Hans E Bøtker, MD, DMSc, Study Director — Department of Cardiovascular research, Aarhus University Hospital, Skejby; Kristian A Thygesen, MD, DMSc, Study Chair — Department of Cardiovascular research, Aarhus University Hospital, Aarhus Hospital; Christian J Terkelsen, MD, PhD, Study Chair — Department of Cardiovascular research, Aarhus University Hospital, Skejby
Locations (1):
- Department of Cardiovascular research, Aarhus University Hospital, Skejby, Dk-8200 Aarhus N, Denmark

REFERENCES:
- [Background] De Luca G, Suryapranata H, Zijlstra F, van 't Hof AW, Hoorntje JC, Gosselink AT, Dambrink JH, de Boer MJ; ZWOLLE Myocardial Infarction Study Group. Symptom-onset-to-balloon time and mortality in patients with acute myocardial infarction treated by primary angioplasty. J Am Coll Cardiol. 2003 Sep 17;42(6):991-7. doi: 10.1016/s0735-1097(03)00919-7. PMID 13678918
- [Background] Boersma E; Primary Coronary Angioplasty vs. Thrombolysis Group. Does time matter? A pooled analysis of randomized clinical trials comparing primary percutaneous coronary intervention and in-hospital fibrinolysis in acute myocardial infarction patients. Eur Heart J. 2006 Apr;27(7):779-88. doi: 10.1093/eurheartj/ehi810. Epub 2006 Mar 2. PMID 16513663
- [Background] Magid DJ, Calonge BN, Rumsfeld JS, Canto JG, Frederick PD, Every NR, Barron HV; National Registry of Myocardial Infarction 2 and 3 Investigators. Relation between hospital primary angioplasty volume and mortality for patients with acute MI treated with primary angioplasty vs thrombolytic therapy. JAMA. 2000 Dec 27;284(24):3131-8. doi: 10.1001/jama.284.24.3131. PMID 11135776
- [Background] Terkelsen CJ, Lassen JF, Norgaard BL, Gerdes JC, Poulsen SH, Bendix K, Ankersen JP, Gotzsche LB, Romer FK, Nielsen TT, Andersen HR. Reduction of treatment delay in patients with ST-elevation myocardial infarction: impact of pre-hospital diagnosis and direct referral to primary percutanous coronary intervention. Eur Heart J. 2005 Apr;26(8):770-7. doi: 10.1093/eurheartj/ehi100. Epub 2005 Jan 31. PMID 15684279
- [Background] Braunwald E, Antman EM, Beasley JW, Califf RM, Cheitlin MD, Hochman JS, Jones RH, Kereiakes D, Kupersmith J, Levin TN, Pepine CJ, Schaeffer JW, Smith EE 3rd, Steward DE, Theroux P, Gibbons RJ, Alpert JS, Eagle KA, Faxon DP, Fuster V, Gardner TJ, Gregoratos G, Russell RO, Smith SC Jr. ACC/AHA guidelines for the management of patients with unstable angina and non-ST-segment elevation myocardial infarction: executive summary and recommendations. A report of the American College of Cardiology/American Heart Association task force on practice guidelines (committee on the management of patients with unstable angina). Circulation. 2000 Sep 5;102(10):1193-209. doi: 10.1161/01.cir.102.10.1193. No abstract available. PMID 10973852
- [Background] Bertrand ME, Simoons ML, Fox KA, Wallentin LC, Hamm CW, McFadden E, De Feyter PJ, Specchia G, Ruzyllo W; Task Force on the Management of Acute Coronary Syndromes of the European Society of Cardiology. Management of acute coronary syndromes in patients presenting without persistent ST-segment elevation. Eur Heart J. 2002 Dec;23(23):1809-40. doi: 10.1053/euhj.2002.3385. No abstract available. PMID 12503543
- [Background] Terkelsen CJ, Lassen JF, Norgaard BL, Gerdes JC, Jensen T, Gotzsche LB, Nielsen TT, Andersen HR. Mortality rates in patients with ST-elevation vs. non-ST-elevation acute myocardial infarction: observations from an unselected cohort. Eur Heart J. 2005 Jan;26(1):18-26. doi: 10.1093/eurheartj/ehi002. Epub 2004 Nov 23. PMID 15615795
- [Background] Koyama Y, Hansen PS, Hanratty CG, Nelson GI, Rasmussen HH. Prevalence of coronary occlusion and outcome of an immediate invasive strategy in suspected acute myocardial infarction with and without ST-segment elevation. Am J Cardiol. 2002 Sep 15;90(6):579-84. doi: 10.1016/s0002-9149(02)02559-6. PMID 12231080
- [Background] Spacek R, Widimsky P, Straka Z, Jiresova E, Dvorak J, Polasek R, Karel I, Jirmar R, Lisa L, Budesinsky T, Malek F, Stanka P. Value of first day angiography/angioplasty in evolving Non-ST segment elevation myocardial infarction: an open multicenter randomized trial. The VINO Study. Eur Heart J. 2002 Feb;23(3):230-8. doi: 10.1053/euhj.2001.2735. PMID 11792138
- [Background] Fox KA, Poole-Wilson PA, Henderson RA, Clayton TC, Chamberlain DA, Shaw TR, Wheatley DJ, Pocock SJ; Randomized Intervention Trial of unstable Angina Investigators. Interventional versus conservative treatment for patients with unstable angina or non-ST-elevation myocardial infarction: the British Heart Foundation RITA 3 randomised trial. Randomized Intervention Trial of unstable Angina. Lancet. 2002 Sep 7;360(9335):743-51. doi: 10.1016/s0140-6736(02)09894-x. PMID 12241831
- [Background] Lagerqvist B, Husted S, Kontny F, Stahle E, Swahn E, Wallentin L; Fast Revascularisation during InStability in Coronary artery disease (FRISC-II) Investigators. 5-year outcomes in the FRISC-II randomised trial of an invasive versus a non-invasive strategy in non-ST-elevation acute coronary syndrome: a follow-up study. Lancet. 2006 Sep 16;368(9540):998-1004. doi: 10.1016/S0140-6736(06)69416-6. PMID 16980115
- [Background] de Winter RJ, Windhausen F, Cornel JH, Dunselman PH, Janus CL, Bendermacher PE, Michels HR, Sanders GT, Tijssen JG, Verheugt FW; Invasive versus Conservative Treatment in Unstable Coronary Syndromes (ICTUS) Investigators. Early invasive versus selectively invasive management for acute coronary syndromes. N Engl J Med. 2005 Sep 15;353(11):1095-104. doi: 10.1056/NEJMoa044259. PMID 16162880
- [Background] Boden WE, O'Rourke RA, Crawford MH, Blaustein AS, Deedwania PC, Zoble RG, Wexler LF, Kleiger RE, Pepine CJ, Ferry DR, Chow BK, Lavori PW. Outcomes in patients with acute non-Q-wave myocardial infarction randomly assigned to an invasive as compared with a conservative management strategy. Veterans Affairs Non-Q-Wave Infarction Strategies in Hospital (VANQWISH) Trial Investigators. N Engl J Med. 1998 Jun 18;338(25):1785-92. doi: 10.1056/NEJM199806183382501. PMID 9632444
- [Background] Hoenig MR, Doust JA, Aroney CN, Scott IA. Early invasive versus conservative strategies for unstable angina & non-ST-elevation myocardial infarction in the stent era. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD004815. doi: 10.1002/14651858.CD004815.pub2. PMID 16856061
- [Background] Breeman A, Ottervanger JP, Boersma E, De Luca G. Coronary revascularization for non-ST elevation acute coronary syndrome: state of the art. J Cardiovasc Med (Hagerstown). 2006 Feb;7(2):108-13. doi: 10.2459/01.JCM.0000203185.66608.2f. PMID 16645369
- [Background] Neumann FJ, Kastrati A, Pogatsa-Murray G, Mehilli J, Bollwein H, Bestehorn HP, Schmitt C, Seyfarth M, Dirschinger J, Schomig A. Evaluation of prolonged antithrombotic pretreatment ("cooling-off" strategy) before intervention in patients with unstable coronary syndromes: a randomized controlled trial. JAMA. 2003 Sep 24;290(12):1593-9. doi: 10.1001/jama.290.12.1593. PMID 14506118
- [Background] Mehta SR, Cannon CP, Fox KA, Wallentin L, Boden WE, Spacek R, Widimsky P, McCullough PA, Hunt D, Braunwald E, Yusuf S. Routine vs selective invasive strategies in patients with acute coronary syndromes: a collaborative meta-analysis of randomized trials. JAMA. 2005 Jun 15;293(23):2908-17. doi: 10.1001/jama.293.23.2908. PMID 15956636
- [Background] Sharir T, Germano G, Waechter PB, Kavanagh PB, Areeda JS, Gerlach J, Kang X, Lewin HC, Berman DS. A new algorithm for the quantitation of myocardial perfusion SPECT. II: validation and diagnostic yield. J Nucl Med. 2000 Apr;41(4):720-7. PMID 10768575
- [Background] Germano G, Kavanagh PB, Berman DS. An automatic approach to the analysis, quantitation and review of perfusion and function from myocardial perfusion SPECT images. Int J Card Imaging. 1997 Aug;13(4):337-46. doi: 10.1023/a:1005815206195. PMID 9306148
- [Background] Cannon CP, Battler A, Brindis RG, Cox JL, Ellis SG, Every NR, Flaherty JT, Harrington RA, Krumholz HM, Simoons ML, Van De Werf FJ, Weintraub WS, Mitchell KR, Morrisson SL, Brindis RG, Anderson HV, Cannom DS, Chitwood WR, Cigarroa JE, Collins-Nakai RL, Ellis SG, Gibbons RJ, Grover FL, Heidenreich PA, Khandheria BK, Knoebel SB, Krumholz HL, Malenka DJ, Mark DB, Mckay CR, Passamani ER, Radford MJ, Riner RN, Schwartz JB, Shaw RE, Shemin RJ, Van Fossen DB, Verrier ED, Watkins MW, Phoubandith DR, Furnelli T. American College of Cardiology key data elements and definitions for measuring the clinical management and outcomes of patients with acute coronary syndromes. A report of the American College of Cardiology Task Force on Clinical Data Standards (Acute Coronary Syndromes Writing Committee). J Am Coll Cardiol. 2001 Dec;38(7):2114-30. doi: 10.1016/s0735-1097(01)01702-8. No abstract available. PMID 11738323
- [Background] Kaltoft A, Bottcher M, Nielsen SS, Hansen HH, Terkelsen C, Maeng M, Kristensen J, Thuesen L, Krusell LR, Kristensen SD, Andersen HR, Lassen JF, Rasmussen K, Rehling M, Nielsen TT, Botker HE. Routine thrombectomy in percutaneous coronary intervention for acute ST-segment-elevation myocardial infarction: a randomized, controlled trial. Circulation. 2006 Jul 4;114(1):40-7. doi: 10.1161/CIRCULATIONAHA.105.595660. Epub 2006 Jun 26. PMID 16801464
- [Background] Mahmarian JJ, Pratt CM, Nishimura S, Abreu A, Verani MS. Quantitative adenosine 201Tl single-photon emission computed tomography for the early assessment of patients surviving acute myocardial infarction. Circulation. 1993 Apr;87(4):1197-210. doi: 10.1161/01.cir.87.4.1197. PMID 8462146
- [Background] Yang H, Pu M, Rodriguez D, Underwood D, Griffin BP, Kalahasti V, Thomas JD, Brunken RC. Ischemic and viable myocardium in patients with non-Q-wave or Q-wave myocardial infarction and left ventricular dysfunction: a clinical study using positron emission tomography, echocardiography, and electrocardiography. J Am Coll Cardiol. 2004 Feb 18;43(4):592-8. doi: 10.1016/j.jacc.2003.07.052. PMID 14975469
- [Background] Andersen HR, Nielsen TT, Rasmussen K, Thuesen L, Kelbaek H, Thayssen P, Abildgaard U, Pedersen F, Madsen JK, Grande P, Villadsen AB, Krusell LR, Haghfelt T, Lomholt P, Husted SE, Vigholt E, Kjaergard HK, Mortensen LS; DANAMI-2 Investigators. A comparison of coronary angioplasty with fibrinolytic therapy in acute myocardial infarction. N Engl J Med. 2003 Aug 21;349(8):733-42. doi: 10.1056/NEJMoa025142. PMID 12930925